CLINICAL TRIAL: NCT01459055
Title: Long-term Ten Years Follow-up in Patients Affected With Acrofacial Vitiligo
Brief Title: Long-term Follow-up in Patients Affected With Acrofacial Vitiligo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Irmandade da Santa Casa de Misericordia de Curitiba (Other)
Responsible Party: Principal Investigator, Caio Cesar Silva de Castro, MD, PhD, Irmandade da Santa Casa de Misericordia de Curitiba
Other Study IDs: ACRO01
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acrofacial vitiligo is a clinical form of vitiligo characterized by macules in distal digits, periorificial-facial and ano-genital areas. Vitiligo European Task Force classifies vitiligo as generalized or localized; generalized vitiligo may be further sub-divided into acrofacial, vulgaris and universalis, and localized vitiligo, into segmental and focal. Some authors do not believe that acrofacial is a real vitiligo clinical form, considering it as an initial form of vulgaris vitiligo. The aim of this study is to follow early- diagnosed acrofacial patients during ten years in order to define if these patients will maintain this clinical form or will evolute to a more severe clinical form.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders, aged older than years, able to understand and provide written informed consent and able to allow compliance at the treatment and the requirements of the protocol;
2. Presence of acrofacial vitiligo;
3. Able to comprehend and willing to provide written informed consent in accordance with institutional and regulatory guidelines.

Exclusion Criteria:

1- Subjects assessed as not suitable for the study in the opinion of the investigator

2 -Inability to complete survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both genders affected by acrofacial vitiligo diagnosed by one single dermatologist.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-01 (Estimated); Study Completion 2020-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Caio C Silva de Castro, MD, PhD, Principal Investigator — Irmandade da Santa Casa de Misericórdia de Curitiba
Locations (1):
- Irmandade da Santa Casa de Misericórdia de Curitiba, Curitiba, Paraná, Brazil